CLINICAL TRIAL: NCT03948711
Title: Brain Oxygenation During Prehospital Anesthesia: an Observational Pilot Study
Brief Title: Brain Oxygenation During Prehospital Anesthesia
Acronym: BOPRA-P
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Oulu University Hospital (Other); FinnHEMS (Unknown)
Responsible Party: Principal Investigator, Jouni Nurmi, MD, senior HEMS physician, associate professor, Helsinki University Central Hospital
Other Study IDs: BOPRA-P
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Near-infrared spectroscopy (NIRS) monitoring of cerebral oxygenation — Monitoring before anesthesia to hospital admission. No treatment decisions made based on monitoring.

SUMMARY:
The study will evaluate the feasibility of Nonin SenSmart H500 device to measuring brain oxygenation during prehospital anesthesia of adult patient. The study also estimates the incidence of cerebral hypoxic events of anesthetized patients during prehospital care. The study does not affect the treatment of the patient. The study is pilot study and will be followed with a main study to assess the association between cerebral oxygenation during prehospital care and outcome of the patient.

ELIGIBILITY:
Inclusion Criteria:

* sedation or anesthesia provided to facilitate endotracheal intubation, performed by HEMS team regardless of the reason

Exclusion Criteria:

* Cardiac arrest at the time of intubation
* Physical barrier for NIRS measuring (e.g. forehead laceration)
* HEMS physician does not escort patient to the hospital (and patient is not dead on the scene after inclusion)
* Workload too high to ensure standard level of clinical care during the study
* Known special vulnerability including known mental disability (permanent, not related to acute condition), patients in nursing homes, prisoners and forensic psychiatric patients.
* Known or evident pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill or trauma patients undergoing prehospital anesthesia and endotracheal intubation for any reason by helicopter emergency medical team providing critical care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Disturbance-free time of the total monitoring time | Prehospital phase
  Proportion of time with readable monitor signal of the total time monitor connected to the patient
Cerebral desaturation events | During prehospital phase after induction of anesthesia
  Number of patients with forehead regional oxygen saturation ≤50% for ≥5 minutes

SECONDARY OUTCOMES:
On-scene time | Prehospital phase
  Time from arrival of helicopter emergency medical services unit on the patient to beginning of transportation
Qualitative feedback from HEMS crews | Prehospital phase
  Comments on the usability of the study device
Survival | 30 days, 12 months
  Data from population registry center
Neurologic disability | 30 days, 12 months
  3-6 on modified Rankin scale (range from 0 [no symptoms at all] to 6 [dead], evaluated by trained research nurse
Health related quality of life | 12 months
  total score of 15-D questionnaire including 15 dimensions each ranked from 1 (good quality of life) to 5 (poor quality of life)

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - FinnHEMS 50 / Oulu University Hospital, Oulu
  - FinnHEMS 10 / Helsinki Univeristy Hospital, Vantaa

IPD SHARING:
Plan to Share IPD: No